CLINICAL TRIAL: NCT00857389
Title: Thiotepa-Clofarabine-Busulfan With Allogeneic Stem Cell Transplant for High Risk Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0363; NCI-2012-01630 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Stem Cell Transplantation; Leukemia; Lymphoma
Keywords: Cancer; Blood And Marrow Transplantation; Stem Cell; Leukemia; Lymphoma; Pediatrics; Bone marrow; Lymph node system; Allogeneic Stem Cell Transplant; ASCT; Busulfan; Busulfex; Myleran; Clofarabine; Clofarex; Clolar; Thiotepa; Antithymocyte globulin; ATG; Thymoglobulin; G-CSF; Filgrastim; Neupogen; Cyclophosphamide; Cytoxan; Neosar; Mesna; Mesnex; Tacrolimus; Prograf; Methotrexate
MeSH Terms: conditions — Leukemia; Lymphoma; Neoplasms | interventions — Thiotepa; Acetyl-CoA C-Acyltransferase; Clofarabine; Hypochlorous Acid; Busulfan; thymoglobulin; Antilymphocyte Serum; Granulocyte Colony-Stimulating Factor; Filgrastim; Tacrolimus; Methotrexate; Cyclophosphamide; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Thio-Clo-Bu with Allo SCT (Experimental): Pre-transplant conditioning regimen:
  Thiotepa (Thio) + Clofarabine (Clo) + Busulfan (Blu) + Allogeneic Stem Cell Transplantation (Allo SCT) + ATG + G-CSF
  Post haploidentical stem cell transplant participants:
  Cyclophosphamide 50 mg/kg by vein on Days + 3 and + 4. Mesna 10 mg/kg by vein just prior to the first dose of cyclophosphamide, repeated every 4 hours for a total of ten (10) doses.
  Interventions: Drug: Thiotepa; Drug: Clofarabine; Drug: Busulfan; Procedure: Allogeneic Stem Cell Transplantation; Drug: Thymoglobulin (ATG); Drug: G-CSF (Filgrastim); Drug: Tacrolimus; Drug: Methotrexate; Drug: Cyclophosphamide; Drug: Mesna

INTERVENTIONS:
Drug: Thiotepa — 5 mg/kg through a central venous catheter (CVC) over 2 hours on Day -8.
  Other Names: Thio
Drug: Clofarabine — 40 mg/m^2 through a central venous catheter (CVC) over 1 hour daily on 4 consecutive days (Days -6 through -3).
  Other Names: Clo; Clofarex; Clolar
Drug: Busulfan — Test dose of 0.5 mg/kg through a central venous catheter (CVC)over 30 minutes on Day -7.
  High dose 5,000 µMol-min through a central venous catheter (CVC) over 3 hours on Days -5, -4, and -3.
  Other Names: Busulfex; Myleran
Procedure: Allogeneic Stem Cell Transplantation — Infusion of stem cells through through a central venous catheter (CVC) On Day 0.
  Other Names: ASCT; SCT
Drug: Thymoglobulin (ATG) — 1.25 mg/kg by vein on Day -4 and 1.75 mg/kg on Day -3.
  Other Names: Antithymocyte globulin
Drug: G-CSF (Filgrastim) — 5 µg/kg Injection under the skin once a day, starting 1 week after transplant, until blood cell levels return to normal.
  Other Names: Neupogen
Drug: Tacrolimus — Starting dose of 0.015 mg/kg (ideal body weight) as a 24 hour continuous infusion daily, to be changed to oral dosing when tolerated. Tacrolimus is to be tapered as indicated after transplant day 90, if no GVHD is present. Tacrolimus is adjusted trough level of 5-15 ng/mL.
  Other Names: Prograf
Drug: Methotrexate — 5 mg/m2 by vein on Days 1, 3 and 6 and Day +11 post transplant. The Day 11 methotrexate dose may be held as indicated if mucositis is present.
Drug: Cyclophosphamide — Post haploidentical stem cell transplant participants: 50 mg/kg by vein on Days + 3 and + 4.
  Other Names: Cytoxan; Neosar
Drug: Mesna — Post haploidentical stem cell transplant participants: 10 mg/kg by vein just prior to the first dose of cyclophosphamide, repeated every 4 hours for a total of ten (10) doses.
  Other Names: Mesnex

SUMMARY:
Any time the words "you," "your," "I," or "me" appear, it is meant to apply to the potential participant.

The goal of this clinical research study is to learn if thiotepa, busulfan, and clofarabine, when given before an allogeneic (bone marrow , blood, or cord blood cells) or haploidentical (bone marrow) stem cell transplantation can help to control cancers of the bone marrow and lymph node system. The safety of this treatment will also be studied.

This is an investigational study. Thiotepa and clofarabine are FDA approved and commercially available for the treatment of leukemia. Busulfan is FDA approved and commercially available for use in stem cell transplantation. The combination of thiotepa, clofarabine, and busulfan together with a stem cell transplant is investigational.

Up to 60 participants will take part in this study. All will be enrolled at M. D. Anderson.

DETAILED DESCRIPTION:
The Study Drugs:

Thiotepa and busulfan are designed to bind to DNA (genetic material of cells), which may cause cancer cells to die. They are commonly used in stem cell transplants.

Clofarabine is designed to interfere with the growth and development of cancer cells.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will begin receiving the study drugs before you receive the stem cell transplant.

The days before you receive your stem cells are called minus days, such as Day -2 and Day -1. The day you receive the stem cells is called Day 0. The days after you receive the stem cells are called plus days, such as Day +1 and Day +2.

On Day -8 (8 days before you receive the stem cell transplant), you will receive thiotepa through a central venous catheter (CVC) over 2 hours. A CVC is a sterile, flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form for this procedure.

On Day -7, you will receive busulfan through a CVC. This dose of busulfan is a low level "test" dose to check how your blood levels change over time. This information will be used to decide the next dose level of busulfan.

Blood (about 1 teaspoon each time) will be drawn 6-11 times total over Days -7 and -5 for pharmacokinetic (PK) testing. PK testing measures the amount of busulfan in the body at different time points. This PK testing will be done to find the dose of busulfan needed for your body size on the other days that you receive busulfan. A heparin lock line will be placed in a vein to lower the number of needed sticks performed for draws. If you cannot have the blood level tests performed for any reason, you will receive the standard busulfan dose.

On Days -6, -5, -4, and -3, you will receive clofarabine through a CVC over 1 hour.

On Days -5, -4, and -3, you will receive busulfan through a CVC over 3 hours.

If you will receive stem cells from a donor whose cells do not match your own cells closely, on Days -4 and -3 you will also receive antithymocyte globulin (ATG) by vein over 4 hours. This will help to reduce the risk of your body rejecting the transplant. If your transplant will involve haploidentical stem cells, you will not receive ATG on Days -4 and -3.

On Days -2 and -1, you will "rest," which means you will not be given any drugs, but your CVC will remain in place.

If thiotepa is not available:

If thiotepa is not available, or if you doctor thinks it is in your best interest, you will receive the following study drugs and total body irradiation (TBI) before you receive the stem cell transplant. TBI involves the delivery of high doses of radiation designed to destroy cancer cells and/or lower the immune system in order to lower the risk of the body rejecting the new stem cells.

Between Days -16 and -7, you will receive a low-level "test" dose of busulfan by vein over about 45 minutes to 1 hour. Test doses are used to study how your body breaks down busulfan and decide the dose of busulfan that you will receive. You may receive the test dose before Day -6 as an outpatient in the clinic, or on Day -6 as an inpatient in the hospital.

Blood (about 1 teaspoon each time) will then be drawn for PK testing up to 11 times over the 11 hours after the busulfan test dose and on Day -4. PK testing measures the amount of study drug in the body at different time points. The study staff will tell you more about the PK testing schedule.

A heparin lock line will be placed in your vein before the PK testing to lower the number of needle sticks needed for these draws. If for any reason it is not possible for the PK tests to be performed, you will receive the standard dose of busulfan.

On Day -7 or Day -6, you will be admitted to the hospital and given fluids through a CVC to hydrate you.

On Days -5, -4, -3, and -2, you will receive clofarabine through a CVC over 1 hour.

On Days -4, -3, and -2, you will receive busulfan through a CVC over 3 hours.

If you will receive stem cells from a donor whose cells do not match your own cells closely, on Days -3 and -2 you will also receive antithymocyte globulin (ATG) by vein over 4 hours. This will help to reduce the risk of your body rejecting the transplant. If your transplant will involve haploidentical stem cells, you will not receive ATG on Days -3 and -2.

On Day -1, you will receive TBI one time.

Stem Cell Transplant:

On Day 0, you will have an allogeneic or haploidentical stem cell transplant through the CVC. Allogeneic stem cells come from a donor whose cells closely match your own cells. Haploidentical stem cells come from a donor whose cells do not match your own cells as closely, but they are specially processed to help prevent graft versus host disease (GVHD).

Receiving stem cells is similar to receiving a blood transfusion. The time required to receive the stem cells will depend on the type of cells you are receiving. Receiving cord blood stem cells can take several minutes. Receiving bone marrow and blood stem cells may take several hours.

You will receive G-CSF (filgrastim) (which helps to produce white blood cells) as an injection under the skin once a day, starting 1 week after the transplant, until your blood cell levels return to normal.

You will receive drugs (mycophenolate mofetil (MMF), tacrolimus and/or methotrexate) to help prevent side effects, such as GVHD. You will receive methylprednisolone if you develop GVHD.

You will stay in the hospital for about 4 weeks after the stem cell transplantation.

If you had a haploidentical stem cell transplant, on Days 3 and 4 after your stem cell transplant, you will receive cyclophosphamide through a CVC over 3 hours. Mesna will be given by vein at the same time you are given each dose of cyclophosphamide, to help protect your bladder from bleeding.

Study Visits:

Beginning on Day -9, once a day while you are in the hospital:

* You will have a physical exam, including measurements of your vital signs.
* You will be asked if you have had any side effects.
* Blood (about 4 tablespoons) will be drawn to test your blood cell counts. Two (2) times a week, this blood will be also be used for routine tests.

After you are out of the hospital, 2 times a month until it has been 100 days after the transplant:

* You will have a physical exam, including measurements of your vital signs and weight.
* You will be asked if you have had any side effects.
* Blood (about 4 tablespoons) will be drawn for routine tests.

About 1, 3, 6, and 12 months after the transplant, blood (about 4 tablespoons) will be drawn to check the status of the disease. You will also have bone marrow aspirations to check the status of the disease. You will also have a physical exam.

If the doctor thinks it is necessary, you may have extra tests and procedures.

Length of Study:

You will be on study for about 1 year. You will be taken off study if the disease gets worse or needs further treatment.

Follow-Up:

If you live close to M. D. Anderson, you will return to the clinical once every several months for a physical exam. At these visits, blood (about 3 teaspoons) will be drawn for routine tests.

You and/or your local doctor will be called every several months and asked about your health status and if the leukemia or MDS has come back.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with one of the following diseases:
2. Acute myelogenous leukemia (AML) in induction failure, relapse, past first remission, or CR1 considered at risk for relapse
3. Myelodysplastic syndromes with International Prognostic Scoring System score (IPSS score) >/= 2 or myelodysplasia that has not responded to chemotherapy
4. Biphenotypic leukemia
5. Acute lymphocytic leukemia with induction failure, first complete remission with high risk cytogenetics (e.g. Philadelphia positive chromosome, t(4:11) Remission requiring more than 2 chemotherapy to achieve remission, or any stage beyond CR1
6. Chronic Myelogenous Leukemia (CML): second chronic phase, accelerated phase or blast crises with less than 10% blasts in the bone marrow, or CR1 and resistance to Gleevec or other tyrosine kinase inhibitors
7. Non-Hodgkin's Lymphoma - induction failures, second or third complete remission, or relapse (including relapse post autologous hematopoietic stem cell transplant)
8. Hodgkin's disease - induction failure, second or later complete remission, or relapse (including relapse post autologous hematopoietic stem cell transplant).
9. Chronic Lymphocytic Leukemia that has failed induction therapy or Rai Stages 2-4
10. Related or unrelated donor which is HLA-matched or mismatched in 1 HLA A, B, C, DR, or DQ locus is acceptable (i.e. >/= 9/10 matched related or unrelated donor, matched with molecular high-resolution technique per current std. for BMT program). Cord blood units must match patient at 4, 5, or 6/6 HLA class 1 serological & II molecular antigens with a min. of 2 x 10e7 TNC/kg recipient weight in the pre-thawed fraction. For patient lacking a matched related or unrelated donor or acceptable cord blood unit(s), a related haploidentical donor (</= 7/8 allele matched at A, B, C, DR loci) may be used.
11. Age </= 60 years.
12. Lansky performance score >/= 50% for patients </= 16 years of age, or Zubrod performance status score of 0-2 for patients > 16 years of age.
13. Cardiac function - left ventricular ejection fraction >/= 40%.
14. Pulmonary function - diffusion capacity of at least 50% predicted. Children unable to perform pulmonary function tests (e.g. less than 7 years old) pulse oximetry of >/= 92% on room air.
15. Serum creatinine < 1.6 mg/dL or creatinine clearance >/= 50 ml/min.
16. SGPT </= 200 IU/mL, serum bilirubin < 1.5 x normal.
17. Written informed consent and assent as is age appropriate.
18. No active infection.

Exclusion Criteria:

1. Pregnancy in women of child bearing potential (pregnancy test performed within 2 weeks of study entry).
2. HIV positive (highly immunosuppressive treatment)
3. Active CNS leukemia
4. Chronic or active Hepatitis B or Hepatitis C. If questions about liver health discuss with PI and strongly consider liver biopsy.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03-02 (Actual); Primary Completion 2019-03-09 (Actual); Study Completion 2019-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kris M. Mahadeo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study received IRB approval October 1, 2008 and was opened to recruitment March 2, 2009. The study remained open to recruitment until August 4, 2015. The study was terminated by the local IRB on April 09, 2019.
Pre-assignment Details: Of the 60 participants enrolled, 2 participants did not proceed to transplant no data were collected for those two participants
Groups:
- Conditioning Reg- Thiotepa, Busulfan, and Clofarabine: Single arm study
Period: Overall Study
Arm/Group | Conditioning Reg- Thiotepa, Busulfan, and Clofarabine
Started | 60
Completed | 58
Not Completed | 2
Not completed — Did not proceed to transplant | 2

BASELINE CHARACTERISTICS:
Population: Two participants did not proceed to transplant no data were collected for those two participants
Groups:
- Conditioning Reg- Thiotepa, Busulfan, and Clofarabine: The 5 mg/kg over 1 hr. Busulfan was administered x 3 days over 3 hr to a daily AUC of 5,000 mcMol-min +/-10%. Clofarabine 40mg/m2 was infused over 1 hr daily x 4 days
Arm/Group | Conditioning Reg- Thiotepa, Busulfan, and Clofarabine
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24
  Between 18 and 65 years | 34
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 25
  More than one race | 0
  Unknown or Not Reported | 21
Region of Enrollment [Number; unit: participants]
  United States | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Survival Rate at 100 Days Post-transplant
Description: The toxicities will be monitored and scored on a daily basis following the methods of Simon R. Practical Bayesian Guideline for Phase IIB Clinical Trials. A Bayesian stopping rule will be used to stop the trial if there is a 90% chance that the true toxicity rate exceeds the target toxicity rate of 0.25.
Time Frame: 100 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Conditioning Reg- Thiotepa, Busulfan, and Clofarabine
Number analyzed (Participants) | 58
Participants | 45

2. Secondary Outcome: Number of Participants With Disease Free Survival
Description: Kaplan-Meier product limit method to estimate the disease free survival.
Time Frame: Up to 2 years post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Conditioning Reg- Thiotepa, Busulfan, and Clofarabine
Number analyzed (Participants) | 58
Participants | 32

3. Secondary Outcome: Overall Survival Rate
Description: Overall Survival Rate will be estimated using the Kaplan-Meier method.
Time Frame: Up to 3 years post transplant
Measure: Median (Full Range); unit: days
Arm/Group | Conditioning Reg- Thiotepa, Busulfan, and Clofarabine
Number analyzed (Participants) | 58
days | 320 [120 to 833]

4. Secondary Outcome: Graft vs Host Disease (GVHD)
Description: Severity of toxicities graded according to the NCI Common Toxicity Criteria Adverse Effects (CTCAE) v3.0. Standard reporting guidelines followed for adverse events. Safety data summarized by category, severity and frequency.
Time Frame: Up to 30 days post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Conditioning Reg- Thiotepa, Busulfan, and Clofarabine
Number analyzed (Participants) | 58
Participants | 34

5. Secondary Outcome: Engraftment
Description: Engraftment is most commonly defined as the first of three consecutive days of achieving a sustained peripheral blood neutrophil count of >500 × 10^6/L .
Time Frame: up to 100 days post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Conditioning Reg- Thiotepa, Busulfan, and Clofarabine
Number analyzed (Participants) | 58
Participants | 52

6. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: as for outcome 4
Time Frame: up to 30 days post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Conditioning Reg- Thiotepa, Busulfan, and Clofarabine
Number analyzed (Participants) | 58
Participants | 52

7. Secondary Outcome: Relapse Rate of Participants Treated With Thiotepa, Busulfan, and Clofarabine
Description: Relapse Rate will be estimated using the Kaplan-Meier method.
Time Frame: Up to 2 years post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Conditioning Reg- Thiotepa, Busulfan, and Clofarabine
Number analyzed (Participants) | 58
Participants | 26

ADVERSE EVENTS:
Time Frame: Adverse events that were related to the preparative regimen and stem cell infusion unil 30 days post transplant.
Arm/Group | Conditioning Reg- Thiotepa, Busulfan, and Clofarabine
All-Cause Mortality (participants affected / at risk) | 16/58
Serious Adverse Events (participants affected / at risk) | 52/58
Other Adverse Events (participants affected / at risk) | 57/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conditioning Reg- Thiotepa, Busulfan, and Clofarabine (N=58)
ARDS- Acute respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 30
Ejection fraction decreased (Cardiac disorders) | 1
DAH-diffuse alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3
ALK increase (Investigations) | 2
Allergic reaction (Immune system disorders) | 2
ALT increase (Investigations) | 12
Hydrocephalus (Nervous system disorders) | 1
Creatinine Increased (Investigations) | 5
Headache (Nervous system disorders) | 1
Hemorrhagic Cystitis (Renal and urinary disorders) | 10
Low granulocyte (Blood and lymphatic system disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
T bilirubin increased (Investigations) | 6
VOD (Hepatobiliary disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 15
Encephalopathy (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conditioning Reg- Thiotepa, Busulfan, and Clofarabine (N=58)
Abodominal Pain (Gastrointestinal disorders) | 3
ALK increased (Investigations) | 10
ALT increase (Investigations) | 18
AMS- altered mental status (Nervous system disorders) | 2
Bleeding (Blood and lymphatic system disorders) | 1
Blurred Vision (Eye disorders) | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 5
Broncholitis Obliterans (Respiratory, thoracic and mediastinal disorders) | 2
Cardiomyopathy (Cardiac disorders) | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1
Confusion (Nervous system disorders) | 1
Creatinine Increased (Investigations) | 9
Cystitis noninfective (Renal and urinary disorders) | 1
DAH-diffuse alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 44
Diplopia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Dry eye (Eye disorders) | 5
Ejection fraction decreased (Cardiac disorders) | 2
Dysrhythmia (Cardiac disorders) | 1
Fever (General disorders) | 22
Flu like symdrome (Musculoskeletal and connective tissue disorders) | 1
Fluid overload (General disorders) | 22
Gastrointestinal bleeding (Gastrointestinal disorders) | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hallucination (Psychiatric disorders) | 1
Hand Foot syndrom (Skin and subcutaneous tissue disorders) | 3
Headache (Nervous system disorders) | 10
Hematochezia (Gastrointestinal disorders) | 1
Hemorrhagic Cystitis (Renal and urinary disorders) | 14
HSCT related microangiopathy (TA-TMA) (Blood and lymphatic system disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 8
Hypotension (Vascular disorders) | 2
Infection (Infections and infestations) | 53
Low platelet (Investigations) | 2
Lower GI track obstruction (Gastrointestinal disorders) | 2
Neuropathy (Nervous system disorders) | 3
Oral mucositis (Gastrointestinal disorders) | 49
Pericarditis (Cardiac disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8
Pruritis (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 23
Secondary graft failure (Blood and lymphatic system disorders) | 3
Seizure (Nervous system disorders) | 3
SK OTH (Skin and subcutaneous tissue disorders) | 1
T bilirubin increased (Investigations) | 14
Nausea (Gastrointestinal disorders) | 57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT00857389/Prot_SAP_000.pdf